CLINICAL TRIAL: NCT04085445
Title: Agent DCB Registry
Brief Title: An "All-Comers" Study of the AgentTM MONORAILTM Paclitaxel-Coated PTCA Balloon Catheter Used in Real-World Clinical Practice in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2460
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chinese Patients Treated With Agent DCB
Keywords: Agent DCB

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: AgentTM MONORAILTM Paclitaxel-Coated PTCA Balloon Catheter — To compile the real-world clinical outcome data for the AgentTM MONORAILTM Paclitaxel-Coated PTCA Balloon Catheter (Agent DCB) used in percutaneous coronary intervention (PCI) in Chinese patients.

SUMMARY:
To compile the real-world clinical outcome data for the AgentTM MONORAILTM Paclitaxel-Coated PTCA Balloon Catheter (Agent DCB) used in percutaneous coronary intervention (PCI) in Chinese patients.

DETAILED DESCRIPTION:
The Agent DCB Registry study will enroll 500 subjects at up to 10 investigational sites in Taiwan, Hong-Kong and Singapore.

If participants decide to participate in this study, participants will first be asked to sign and date this consent form. If participants sign the consent form, participants will go through a baseline/ procedure process. Information about participants and participants' health will be collected and participants will have a limited physical examination.

Participants will need to have the laboratory tests (including myocardial enzyme test before and post the index procedure, pregnancy test before the index procedure) and other assessments to find out if participants meet the requirements to be in the study and to ensure it is safe for participants to have the procedure. These tests and assessments are part of routine care and may be done even if participants do not join the study. If participants have had some of them recently, they may not need to be repeated.

Participants will be expected to follow the scheduled follow-ups which occur at 30 days, 6 and 12 months, and then annually through 3 years post the index procedure for all enrolled subjects. Angiographic follow-up will perform at 9 months post index procedure for all the subjects with small vessel lesions and the first 100 consecutively enrolled subjects with ISR lesions. Enrolled subjects with the failure of advancing Agent DCB across target lesion will be followed through hospital discharge following the initial attempted index procedure.

Participants' participation in the study will be completed after approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subject at least 18 years of age(or meet age requirements per local law).
* Subject (or legal guardian) who understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
* Subject who has ischemic symptoms or evidence of myocardial ischemia and is clinically indicated for PCI and will be treated with Agent DCB.
* Subject is willing to comply with all protocol-required follow-up evaluation.
* In women with childbearing potential a negative pregnancy test is mandatory.
* Subject with no known intolerance to paclitaxel and no contraindications to antiplatelet regimen.

Exclusion Criteria:

- Exclusion criteria are not required in the Agent DCB registry study as it is an "all comers" study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All enrolled subjects will be eligible for evaluation. The inclusion and exclusion criteria for the Agent DCB Registry study are listed in the following sections.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with 12 months post index procedure | 12 months
  Major adverse cardiac event (MACE) rate, defined as cardiac death, myocardial infarction (MI, Q-wave and non-Q-wave) and target vessel revascularization (TVR),Target lesion revascularization (TLR) and target lesion failure (TLF) rates

CONTACTS AND LOCATIONS:
Locations (9):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Tan Tock Seng Hospital, Singapore, Singapore
- Taiwan (7):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Cheng Hsin General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided